CLINICAL TRIAL: NCT05907499
Title: Low Dose Decitabine for Poor Graft Function Post Allogenic Hematopoietic Stem Cell Transplantation
Brief Title: Decitabine for Poor Graft Function Post Allo-HSCT
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOOCHOW-HY-2023-06-06
Record Dates: First submitted 2023-06-08; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Poor Graft Function
Keywords: poor graft function; hematopoietic stem cell transplantation
MeSH Terms: interventions — Decitabine; Granulocyte Colony-Stimulating Factor; eltrombopag; avatrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Decitabine 6 mg/m2 daily subcutaneously for consecutive 3 days (day 1 to day 3)
  Interventions: Drug: Decitabine; Drug: Granulocyte Colony-Stimulating Factor; Drug: Thrombopoietin Receptor Agonist; Drug: Recombinant human erythropoietin
- Arm B (Active Comparator): The hematologic growth factors (granulocyte-colony stimulating factor, thrombopoietin receptor agonists, recombinant human erythropoietin)
  Interventions: Drug: Granulocyte Colony-Stimulating Factor; Drug: Thrombopoietin Receptor Agonist; Drug: Recombinant human erythropoietin

INTERVENTIONS:
Drug: Decitabine — Decitabine 6 mg/m2 daily subcutaneously for consecutive 3 days (day 1 to day 3)
  Other Names: Dec
  Arms: Arm A
Drug: Granulocyte Colony-Stimulating Factor — 5ug/kg/d when absolute neutrophil count ≤ 1.5 × 109/L
  Other Names: G-CSF
Drug: Thrombopoietin Receptor Agonist — Eltrombopag initial dose: 25 mg orally once a day, may increase to up to 75 mg/day, when platelet count ≤ 30 × 109/L; Avatrombopag initial dose: 20 mg orally once a day, may increase to up to 60 mg/day, when platelet count ≤ 30 × 109/L.
  Other Names: Eltrombopag / Avatrombopag
Drug: Recombinant human erythropoietin — 10000 U/day when hemoglobin ≤ 85 g/L
  Other Names: EPO

SUMMARY:
This randomized trial aims at validating the efficacy and safety of low-dose decitabine for PGF post allo-HSCT.

DETAILED DESCRIPTION:
Poor graft function (PGF), defined by the presence of multilineage cytopenias in the presence of 100% donor chimerism, is a serious complication of allogeneic stem cell transplant (allo-HSCT). Emerging evidence demonstrates that the inadequate stem cells infusion, bone marrow microenvironment and immune dysregulation play a crucial role in maintaining and regulating hematopoiesis. Current therapies remain debatable, including selected CD34+ cells infusion, mesenchymal stromal cells infusion, prophylactic N-acetyl cysteine administration, etc. Thereafter, the investigators conduct a randomized trial aiming at validating the efficacy and safety of low-dose decitabine in PGF post allo-HSCT patients.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed as PGF at day 28 post-HSCT or later. PGF was defined as two or three cytopenias, absolute neutrophil count ≤ 1.5 × 109/L, platelet count ≤ 30 × 109/L, hemoglobin ≤ 85g/L, lasting for more than 2 consecutive weeks;
2. Full donor chimerism;
3. Primary disease in remission;
4. No severe GVHD and relapse;
5. ECOG: 0-2;
6. Expected survival longer than 1 month

Exclusion Criteria:

1. Allergic to decitabine;
2. Active infections;
3. Uncontrolled GVHD;
4. Severe organ dysfunction;
5. Relapse of underlying malignancies;
6. Graft failure;
7. Received decitabine or participated in other clinical trials within one month before screening.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
The treatment response | day +28
  The rate of hematological response of after HSCT
Survival | 1 year
  The rate of overall survival

SECONDARY OUTCOMES:
Bone marrow recovery | day +28
  Number of participants with granulopoiesis, erythropoiesis and megakaryopoiesis recovery of bone marrow after HSCT
Relapse and GVHD | 3-month
  The rate of relapse and GVHD after HSCT
Event free survival | 1 year
  The rate of event free survival after HSCT

CONTACTS AND LOCATIONS:
Overall Officials: Yue Han, Professor, Principal Investigator — The First Affiliated Hospital of Soochow University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alchalby H, Yunus DR, Zabelina T, Ayuk F, Kroger N. Incidence and risk factors of poor graft function after allogeneic stem cell transplantation for myelofibrosis. Bone Marrow Transplant. 2016 Sep;51(9):1223-7. doi: 10.1038/bmt.2016.98. Epub 2016 Apr 18. PMID 27088376
- [Background] Larocca A, Piaggio G, Podesta M, Pitto A, Bruno B, Di Grazia C, Gualandi F, Occhini D, Raiola AM, Dominietto A, Bregante S, Lamparelli T, Tedone E, Oneto R, Frassoni F, Van Lint MT, Pogliani E, Bacigalupo A. Boost of CD34+-selected peripheral blood cells without further conditioning in patients with poor graft function following allogeneic stem cell transplantation. Haematologica. 2006 Jul;91(7):935-40. PMID 16818281
- [Background] Prabahran A, Koldej R, Chee L, Ritchie D. Clinical features, pathophysiology, and therapy of poor graft function post-allogeneic stem cell transplantation. Blood Adv. 2022 Mar 22;6(6):1947-1959. doi: 10.1182/bloodadvances.2021004537. PMID 34492685
- [Background] Ghobadi A, Fiala MA, Ramsingh G, Gao F, Abboud CN, Stockerl-Goldstein K, Uy GL, Grossman BJ, Westervelt P, DiPersio JF. Fresh or Cryopreserved CD34+-Selected Mobilized Peripheral Blood Stem and Progenitor Cells for the Treatment of Poor Graft Function after Allogeneic Hematopoietic Cell Transplantation. Biol Blood Marrow Transplant. 2017 Jul;23(7):1072-1077. doi: 10.1016/j.bbmt.2017.03.019. Epub 2017 Mar 18. PMID 28323004
- [Background] Lubbert M, Suciu S, Baila L, Ruter BH, Platzbecker U, Giagounidis A, Selleslag D, Labar B, Germing U, Salih HR, Beeldens F, Muus P, Pfluger KH, Coens C, Hagemeijer A, Eckart Schaefer H, Ganser A, Aul C, de Witte T, Wijermans PW. Low-dose decitabine versus best supportive care in elderly patients with intermediate- or high-risk myelodysplastic syndrome (MDS) ineligible for intensive chemotherapy: final results of the randomized phase III study of the European Organisation for Research and Treatment of Cancer Leukemia Group and the German MDS Study Group. J Clin Oncol. 2011 May 20;29(15):1987-96. doi: 10.1200/JCO.2010.30.9245. Epub 2011 Apr 11. PMID 21483003
- [Background] Han P, Yu T, Hou Y, Zhao Y, Liu Y, Sun Y, Wang H, Xu P, Li G, Sun T, Hu X, Liu X, Li L, Peng J, Zhou H, Hou M. Low-Dose Decitabine Inhibits Cytotoxic T Lymphocytes-Mediated Platelet Destruction via Modulating PD-1 Methylation in Immune Thrombocytopenia. Front Immunol. 2021 Feb 17;12:630693. doi: 10.3389/fimmu.2021.630693. eCollection 2021. PMID 33679776
- [Background] Han P, Hou Y, Zhao Y, Liu Y, Yu T, Sun Y, Wang H, Xu P, Li G, Sun T, Hu X, Liu X, Li L, Peng J, Zhou H, Hou M. Low-dose decitabine modulates T-cell homeostasis and restores immune tolerance in immune thrombocytopenia. Blood. 2021 Aug 26;138(8):674-688. doi: 10.1182/blood.2020008477. PMID 33876188
- [Background] Zambuzi FA, Cardoso-Silva PM, Castro RC, Fontanari C, Emery FDS, Frantz FG. Decitabine Promotes Modulation in Phenotype and Function of Monocytes and Macrophages That Drive Immune Response Regulation. Cells. 2021 Apr 12;10(4):868. doi: 10.3390/cells10040868. PMID 33921194
- [Background] Kopp LM, Ray A, Denman CJ, Senyukov VS, Somanchi SS, Zhu S, Lee DA. Decitabine has a biphasic effect on natural killer cell viability, phenotype, and function under proliferative conditions. Mol Immunol. 2013 Jul;54(3-4):296-301. doi: 10.1016/j.molimm.2012.12.012. Epub 2013 Jan 16. PMID 23328088
- [Background] Tang Y, Chen J, Liu Q, Chu T, Pan T, Liang J, He XF, Chen F, Yang T, Ma X, Wu X, Hu S, Cao X, Hu X, Hu J, Liu Y, Qi J, Shen Y, Ruan C, Han Y, Wu D. Low-dose decitabine for refractory prolonged isolated thrombocytopenia after HCT: a randomized multicenter trial. Blood Adv. 2021 Mar 9;5(5):1250-1258. doi: 10.1182/bloodadvances.2020002790. PMID 33646303
- [Background] Han Y, Tang Y, Chen J, Liang J, Ye C, Ruan C, Wu D. Low-Dose Decitabine for Patients With Thrombocytopenia Following Allogeneic Hematopoietic Stem Cell Transplantation: A Pilot Therapeutic Study. JAMA Oncol. 2015 May;1(2):249-51. doi: 10.1001/jamaoncol.2014.316. No abstract available. PMID 26181032
- [Background] DeSimone J, Koshy M, Dorn L, Lavelle D, Bressler L, Molokie R, Talischy N. Maintenance of elevated fetal hemoglobin levels by decitabine during dose interval treatment of sickle cell anemia. Blood. 2002 Jun 1;99(11):3905-8. doi: 10.1182/blood.v99.11.3905. PMID 12010787